CLINICAL TRIAL: NCT06851988
Title: Can Exercise Ameliorate Immunosenescence and Thereby Reduce Relapse in Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jason Chia-Hsun Hsieh, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202201332B0
Record Dates: First submitted 2024-02-21; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Aging; High-intensity Interval Training; Head and Neck Cancers - Tonsils
Keywords: Exercise; Immunosenescence; Recurrence-free survival; Head and Neck Cancer
MeSH Terms: conditions — Motor Activity; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head and Neck patient after CCRT treatment with HIIT training (Experimental): After CCRT treatment 4-5 week arrange HIIT training for patient. Two to three times a week ,total 24-36 times.
  keep follow the PFS and OS
  Interventions: Other: HIIT & Record of physical activities at home.; Other: HIIT only
- Head and Neck patient after CCRT treatment (No Intervention): keep follow the PFS and OS

INTERVENTIONS:
Other: HIIT & Record of physical activities at home. — After CCRT treatment 4-5 week arrange HIIT excise for patient two to three times a week 24-36 times. And record of physical activities at home. According to the record set goal to acheive.
  Arms: Head and Neck patient after CCRT treatment with HIIT training
Other: HIIT only — After CCRT treatment 4-5 week arrange HIIT excise for patient two to three times a week 24-36 times.
  Arms: Head and Neck patient after CCRT treatment with HIIT training

SUMMARY:
Through the implementation of this three-year project, investigators expect to find a safe and effective exercise prescription for patients with oral cancer after surgery. The findings will encourage and promise and add further support to the concept that exercise prescription is worth implementation as part of care for the patients with head and neck cancer.

DETAILED DESCRIPTION:
Cancer patients have theoretically returned to a disease-free state after receiving curative anticancer therapy, but even after receiving adjuvant concurrent chemoradiotherapy, it does not ideally prevent all cancer recurrences. For that, several guidelines recommend that cancer survivors participate in regular exercise. Exercise has been thought to be associated with improved outcomes and mortality in healthy individuals as well as in certain cancer populations. However, the most robust evidence demonstrated in patients with prostate, breast and colorectal cancers, the effectiveness of exercise interventions in Head and Neck cancer survivors is inadequately understood.

Aging of the immune system (so-called immunosenescence) has long been known to increase the risk of infection, cancer, chronic inflammatory diseases and age-related multi-morbidity in humans. In the literatures, patients with oral cavity cancer are also believed to have the phenomenon of immune aging (immunosenescence). One of the mechanisms that maintain cellular homeostasis and prevent immunosenescence-related damage is autophagy, a cell-survival mechanism, and it has been proposed as one of the most powerful antiaging therapies. Regular exercise can reestablish autophagy, probably through AMP-activated protein kinase activation, and help in reducing the age-related senescence diseases. At present, many research teams in cancer centers are trying to design large-scale prospective trials to answer whether the intervention of exercise can avoid cancer occurrence, health promotion in survivors, and prevention of recurrence.

This project focus on the integration of the basic and clinical research. The multidisciplinary research teams include participants of the Department of Hematology and Oncology and Department of Rehabilitation of the New Taipei City Tucheng Hospital. The main purpose of three-year project is to investigate whether high-intensity interval training (HIIT) along with resistance exercise intervention, which could reduce the recurrence rate by ameliorating immunosenescence on patients with head and neck cancer. The main tasks order by year of this project are as the following: (1) investigating the differences of immunosenescence indicators in blood with before and after conducting eight weeks of HIIT along with resistance exercise training for patients with head and neck cancer (1st year plan); (2) recruiting new subjects, gathering the physical activity at home and the cancer recurrence rate for first-year subjects, investigating the differences of immunosenescence indicators and immune indicators in the peripheral blood, and examining the clinical effectiveness of exercise training (2nd year plan); (3) tracking above research materials for subjects including recruiting in the first and second years (3rd year plan). Through the implementation of this three-year project, investigators expect to find a safe and effective exercise prescription for patients with oral cancer after surgery. The findings will encourage and promise and add further support to the concept that exercise prescription is worth implementation as part of care for the patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20
2. Pathology:Squamous cell carcinoma
3. Need CCRT treatment
4. ECOG PS<2
5. Agree with blood drawing, excise training, questionnaire

Exclusion Criteria:

1. ECOG PS≥2
2. Unable to tolerate basic exercise, or CCRT treatment
3. Mental illness or any medical illness or concurrent illness that may be aggravated by exercise training or unmanageable
4. Any medical condition that unsuitable for exercise
5. Disagree to trial procedures: exercise, blood draws, questionnaire

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
% of participants with phenoage and age | 1 month, after CCRT
  To evaluate the phenoage acceleration by calculating differencehe of patients with phenoage and age.
% of participants with phenoage and age | 6 month, after CCRT
  To evaluate the phenoage acceleration by calculating differencehe of patients with phenoage and age.
Peak VO2 (ml/min/kg) of participants | baseline
  To record the Peak VO2 (ml/min/kg) of participants and to evulate the effectiveness of exercise training
Peak VO2 (ml/min/kg) of participants | 1 month, after CCRT
  To record the Peak VO2 (ml/min/kg) of participants and to evulate the effectiveness of exercise training
Peak VO2 (ml/min/kg) of participants | 6 month, after CCRT
  To record the Peak VO2 (ml/min/kg) of participants and to evulate the effectiveness of exercise training
Questionnaire of European Organisation for Research and Treatment of Cancer Quality of Life Head and Neck Module (EORTC QLQ-HN43) | baseline
  To assese the quality of life at the Head and Neck participants and evulate the effectiveness of exercise training.The minimum value is 43 and the maximum value is 172
Questionnaire of European Organisation for Research and Treatment of Cancer Quality of Life Head and Neck Module (EORTC QLQ-HN43) | 1 month, after CCRT
  To assese the quality of life at the Head and Neck participants and evulate the effectiveness of exercise training.The minimum value is 43 and the maximum value is 172
Questionnaire of European Organisation for Research and Treatment of Cancer Quality of Life Head and Neck Module (EORTC QLQ-HN43) | 6 month, after CCRT
  To assese the quality of life at the Head and Neck participants and evulate the effectiveness of exercise training.The minimum value is 43 and the maximum value is 172

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, Study Chair — New Tipei City Tucheng Hospital
Locations (1):
- TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No